CLINICAL TRIAL: NCT06680791
Title: Molecular Classification in Relation to Prevention of Endometrial Cancer Recurrence and Lifestyle Factors
Acronym: MPEC
Status: Recruiting | Type: Observational
Sponsor: Lukas Vanek (Other Government)
Collaborators: National Institute of Public Health (NIPH), Czech Republic (Unknown)
Responsible Party: Sponsor-Investigator, Lukas Vanek, Medical doctor, Department of Gynecology and Obstetrics, Faculty Hospital Kralovske Vinohrady
Organization: Faculty Hospital Kralovske Vinohrady (Other Government)
Other Study IDs: NW24-09-00505
Record Dates: First submitted 2024-06-10; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Endometrial Cancer; Genetic Predisposition; Risk Behavior
Keywords: Endometrial cancer; BMI; Hypertension; Diabetes mellitus; Genetic predispositions
MeSH Terms: conditions — Endometrial Neoplasms; Genetic Predisposition to Disease; Risk-Taking; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients with endometrial cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometrial cancer (EC) is one of the most prevalent cancers in women worldwide with a significantly increasing incidence, especially in developed countries. One of the reasons for the increase in the incidence of this disease is the rising incidence of obesity as the biggest risk factor for the development of this disease. Other important risk factors are hypertension, diabetes mellitus and the general ageing of the population. These risk factors are not only associated with a higher risk of developing the disease, but also, for example, with post-operative complications affecting the quality of life of patients after surgery. The molecular classification of endometrial cancer, which has been introduced into clinical practice in recent years, is currently helping physicians to make treatment decisions for individual patients and predict prognosis. In this project, we would like to focus on the relationship of this molecular classification with genomic mutational signatures detected by whole-exome sequencing and their association with lifestyle risk factors for endometrial cancer (obesity - BMI, hypertension, diabetes mellitus), including the extent of staging lymphadenectomy. Identification and detailed analysis of dominant mutational profiles associated with a specific molecular subtype of EC and their influence on the presence of lifestyle risk factors may have a major impact on both disease development and prevention of disease recurrence. The possible relationship of the mutational profile with the extent of staging lymphadenectomy may help in deciding the extent of this surgical procedure, which subsequently affects the quality of life of patients, especially in patients with high BMI. Given the widespread prevalence of lifestyle risk factors in the developed world, a detailed understanding of the relationship between the genetic profile, its alterations and the prevalence of these risk factors, with potentially major implications for treatment success, is crutial.

DETAILED DESCRIPTION:
The main goal of the project is to define specific mutational signatures of endometrial cancer (EC) patients using whole-exome sequencing technology. The relationship between mutational profiles and molecular classification of endometrial cancer will be analyzed in order to improve the stratification of these patients, especially those classified as having a non-specific molecular profile or p53 mutations. At the same time, the association between the dominant mutational profiles of EC patients with the prevalence of lifestyle risk factors such as obesity/BMI, hypertension and diabetes mellitus will be investigated and their incidence is becoming more prevalent in the modern population. Associations between the occurrence of specific mutation profiles with risk factors will be sought and their role in influencing the genetic profile of EC patients will be analyzed. Another aim of the project is to find relationships between specific mutational profiles of patients with the extent of staging lymphadenectomy, which could help to decide the extent of this surgery, which subsequently affects the quality of life of patients, especially in patients with high BMI. The final aim of the project is to establish a methodology to detect mutations arising from dominant specific mutational profiles in circulating tumor DNA (ctDNA) to monitor potential recurrence in patients at high risk of developing and recurrent disease. Overall, the main contribution of the project will be a detailed understanding of the relationship of the genetic profile of EC patients with their molecular subtype, the extent of staging lymphadenectomy and, most importantly, their impact related to the presence of lifestyle risk factors. These factors may be related to the presence of specific dominant mutational profiles subsequently serving as a tool for prognosis, prevention, risk of recurrence but also potential therapeutic targets in women with the presence of any of the lifestyle risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of endometrial cancer.
* Treated with uterine removal with adequate staging.

Exclusion Criteria:

* There are no exclusion criteria in this study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients surgically treated with hysterectomy in Department of Gynecology and Obstetrics, Faculty hospital Královské Vinohrady.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Genetic variants/mutation signatures | Sampled during surgery
  Association of dominant signatures with molecular subtype, staging lymphadenectomy, age and lifestyle risk factors as well as their role in recurrence prediction of high-risk patients (obese patients, patients with p53 abnormalities, NSMP patients) and for surgical treatment decisions.
Quality of life of EC patients using the EORTC QLQ-C30 questionnaire | Questionnaires filled before surgery, then after 6,12,24 months
  Analysis of endometrial cancer patients' quality of life undergoing hysterectomy with adequate staging lymphadenectomy by questionary study, specifically questionnaire European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30).
  The questionnaire is composed of both multi item scales and single item scales. These include five functional scales, three symptom scales, global health status/quality of life scale and six single items.
  All scales and single item measures range in score from 0 to 100, high scale represents a higher response level - high score for a functional scale represents a high/healthy level of functioning, high score for the global health status/quality of life represents a high quality of life, high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life of EC patients using the EORTC QLQ-EN24 questionnaire | Questionnaires filled before surgery, then after 6,12,24 months
  Analysis of endometrial cancer patients' quality of life undergoing hysterectomy with adequate staging lymphadenectomy by questionary study, specifically questionnaire European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Endometrial Cancer Module (EORTC QLQ-EN24).
  The questionnaire is composed of three functional, single-item scales, and 10 symptom scales (both multi-item scales and single-item measures).
  All scales and single item measures range in score from 0 to 100, high scale represents a higher response level - high score for a functional scale represents a high/healthy level of functioning, high score for a symptom scale/item represents a high level of symptomatology/problems.
Physical activity of EC patients | Questionnaires filled before surgery, then after 6,12,24 months
  Analysis of physical activity of EC patients' undergoing hysterectomy with adequate staging lymphadenectomy by questionary study, specifically International Physical Activity Questionnaire - Short Form (IPAQ-SF) questionnaire. This questionnaire assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting. MET (metabolic equivalent) minutes represent the amount of energy expended carrying out physical activity.
  Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) depending on MET-minutes (higher score means higher category) and sitting time (higher score means lower category).
Introduction of methodology of ctDNA detection by digital PCR of consecutive follow-up samples. | Collection of blood samples at the day of surgery, then after 6,12 and 24 months
  Collection of follow-up blood samples at different time-points, at the day of surgery, and then during 6, 12 and 24 months after surgery, methodology optimization for genetic variant detection in ctDNA isolated from follow-up blood samples, analysis of somatic variants resulting from dominant molecular signatures in ctDNA with potential role in EC progress or recurrence, mainly for high-risk EC patients (patients with p53 abnormal expression and NSMP group).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Halaška, prof. MUDr., Principal Investigator — Medical director
Locations (1):
- Faculty Hospital Královské Vinohrady, Prague, Czechia

REFERENCES:
- [Background] Akesson A, Wolmesjo N, Adok C, Milsom I, Dahm-Kahler P. Lymphadenectomy, obesity and open surgery are associated with surgical complications in endometrial cancer. Eur J Surg Oncol. 2021 Nov;47(11):2907-2914. doi: 10.1016/j.ejso.2021.06.034. Epub 2021 Jul 1. PMID 34238643
- [Background] Alexandrov LB, Kim J, Haradhvala NJ, Huang MN, Tian Ng AW, Wu Y, Boot A, Covington KR, Gordenin DA, Bergstrom EN, Islam SMA, Lopez-Bigas N, Klimczak LJ, McPherson JR, Morganella S, Sabarinathan R, Wheeler DA, Mustonen V; PCAWG Mutational Signatures Working Group; Getz G, Rozen SG, Stratton MR; PCAWG Consortium. The repertoire of mutational signatures in human cancer. Nature. 2020 Feb;578(7793):94-101. doi: 10.1038/s41586-020-1943-3. Epub 2020 Feb 5. PMID 32025018
- [Background] Ashley CW, Da Cruz Paula A, Kumar R, Mandelker D, Pei X, Riaz N, Reis-Filho JS, Weigelt B. Analysis of mutational signatures in primary and metastatic endometrial cancer reveals distinct patterns of DNA repair defects and shifts during tumor progression. Gynecol Oncol. 2019 Jan;152(1):11-19. doi: 10.1016/j.ygyno.2018.10.032. Epub 2018 Nov 8. PMID 30415991
- [Background] Ashley CW, Selenica P, Patel J, Wu M, Nincevic J, Lakhman Y, Zhou Q, Shah RH, Berger MF, Da Cruz Paula A, Brown DN, Marra A, Iasonos A, Momeni-Boroujeni A, Alektiar KM, Long Roche K, Zivanovic O, Mueller JJ, Zamarin D, Broach VA, Sonoda Y, Leitao MM, Friedman CF, Jewell E, Reis-Filho JS, Ellenson LH, Aghajanian C, Abu-Rustum NR, Cadoo K, Weigelt B. High-Sensitivity Mutation Analysis of Cell-Free DNA for Disease Monitoring in Endometrial Cancer. Clin Cancer Res. 2023 Jan 17;29(2):410-421. doi: 10.1158/1078-0432.CCR-22-1134. PMID 36007103
- [Background] Barry JA, Azizia MM, Hardiman PJ. Risk of endometrial, ovarian and breast cancer in women with polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod Update. 2014 Sep-Oct;20(5):748-58. doi: 10.1093/humupd/dmu012. Epub 2014 Mar 30. PMID 24688118
- [Background] Bhaskaran K, Douglas I, Forbes H, dos-Santos-Silva I, Leon DA, Smeeth L. Body-mass index and risk of 22 specific cancers: a population-based cohort study of 5.24 million UK adults. Lancet. 2014 Aug 30;384(9945):755-65. doi: 10.1016/S0140-6736(14)60892-8. Epub 2014 Aug 13. PMID 25129328
- [Background] Bolivar AM, Luthra R, Mehrotra M, Chen W, Barkoh BA, Hu P, Zhang W, Broaddus RR. Targeted next-generation sequencing of endometrial cancer and matched circulating tumor DNA: identification of plasma-based, tumor-associated mutations in early stage patients. Mod Pathol. 2019 Mar;32(3):405-414. doi: 10.1038/s41379-018-0158-8. Epub 2018 Oct 12. PMID 30315273
- [Background] Crosbie EJ, Zwahlen M, Kitchener HC, Egger M, Renehan AG. Body mass index, hormone replacement therapy, and endometrial cancer risk: a meta-analysis. Cancer Epidemiol Biomarkers Prev. 2010 Dec;19(12):3119-30. doi: 10.1158/1055-9965.EPI-10-0832. Epub 2010 Oct 28. PMID 21030602
- [Background] Crosbie EJ, Kitson SJ, McAlpine JN, Mukhopadhyay A, Powell ME, Singh N. Endometrial cancer. Lancet. 2022 Apr 9;399(10333):1412-1428. doi: 10.1016/S0140-6736(22)00323-3. PMID 35397864
- [Background] Fekete JT, Gyorffy B. ROCplot.org: Validating predictive biomarkers of chemotherapy/hormonal therapy/anti-HER2 therapy using transcriptomic data of 3,104 breast cancer patients. Int J Cancer. 2019 Dec 1;145(11):3140-3151. doi: 10.1002/ijc.32369. Epub 2019 May 7. PMID 31020993
- [Background] Grady D, Gebretsadik T, Kerlikowske K, Ernster V, Petitti D. Hormone replacement therapy and endometrial cancer risk: a meta-analysis. Obstet Gynecol. 1995 Feb;85(2):304-13. doi: 10.1016/0029-7844(94)00383-O. PMID 7824251
- [Background] Grant BM, Pugh TJ, Oza AM. Molecular Monitoring in Endometrial Cancer-Ready for Prime Time? Clin Cancer Res. 2023 Jan 17;29(2):305-308. doi: 10.1158/1078-0432.CCR-22-2781. PMID 36354753
- [Background] Gu B, Shang X, Yan M, Li X, Wang W, Wang Q, Zhang C. Variations in incidence and mortality rates of endometrial cancer at the global, regional, and national levels, 1990-2019. Gynecol Oncol. 2021 May;161(2):573-580. doi: 10.1016/j.ygyno.2021.01.036. Epub 2021 Feb 5. PMID 33551200
- [Background] Harris HR, Terry KL. Polycystic ovary syndrome and risk of endometrial, ovarian, and breast cancer: a systematic review. Fertil Res Pract. 2016 Dec 5;2:14. doi: 10.1186/s40738-016-0029-2. eCollection 2016. PMID 28620541
- [Background] Hlavac V, Holy P, Vaclavikova R, Rob L, Hruda M, Mrhalova M, Cernaj P, Bouda J, Soucek P. Whole-exome sequencing of epithelial ovarian carcinomas differing in resistance to platinum therapy. Life Sci Alliance. 2022 Oct 13;5(12):e202201551. doi: 10.26508/lsa.202201551. PMID 36229065
- [Background] Hlavac V, Cervenkova L, Susova S, Holy P, Liska V, Vycital O, Sorejs O, Fiala O, Daum O, Soucek P. Exome Sequencing of Paired Colorectal Carcinomas and Synchronous Liver Metastases for Prognosis and Therapy Prediction. JCO Precis Oncol. 2023 May;7:e2200557. doi: 10.1200/PO.22.00557. PMID 37141551
- [Background] Hubackova S, Pribyl M, Kyjacova L, Moudra A, Dzijak R, Salovska B, Strnad H, Tambor V, Imrichova T, Svec J, Vodicka P, Vaclavikova R, Rob L, Bartek J, Hodny Z. Interferon-regulated suprabasin is essential for stress-induced stem-like cell conversion and therapy resistance of human malignancies. Mol Oncol. 2019 Jul;13(7):1467-1489. doi: 10.1002/1878-0261.12480. Epub 2019 Jun 10. PMID 30919591
- [Background] Jamieson A, Barroilhet LM, McAlpine JN. Molecular classification in endometrial cancer: Opportunities for precision oncology in a changing landscape. Cancer. 2022 Aug 1;128(15):2853-2857. doi: 10.1002/cncr.34328. Epub 2022 Jun 3. PMID 35657171
- [Background] Lai Z, Markovets A, Ahdesmaki M, Chapman B, Hofmann O, McEwen R, Johnson J, Dougherty B, Barrett JC, Dry JR. VarDict: a novel and versatile variant caller for next-generation sequencing in cancer research. Nucleic Acids Res. 2016 Jun 20;44(11):e108. doi: 10.1093/nar/gkw227. Epub 2016 Apr 7. PMID 27060149
- [Background] Lawrence MS, Stojanov P, Polak P, Kryukov GV, Cibulskis K, Sivachenko A, Carter SL, Stewart C, Mermel CH, Roberts SA, Kiezun A, Hammerman PS, McKenna A, Drier Y, Zou L, Ramos AH, Pugh TJ, Stransky N, Helman E, Kim J, Sougnez C, Ambrogio L, Nickerson E, Shefler E, Cortes ML, Auclair D, Saksena G, Voet D, Noble M, DiCara D, Lin P, Lichtenstein L, Heiman DI, Fennell T, Imielinski M, Hernandez B, Hodis E, Baca S, Dulak AM, Lohr J, Landau DA, Wu CJ, Melendez-Zajgla J, Hidalgo-Miranda A, Koren A, McCarroll SA, Mora J, Crompton B, Onofrio R, Parkin M, Winckler W, Ardlie K, Gabriel SB, Roberts CWM, Biegel JA, Stegmaier K, Bass AJ, Garraway LA, Meyerson M, Golub TR, Gordenin DA, Sunyaev S, Lander ES, Getz G. Mutational heterogeneity in cancer and the search for new cancer-associated genes. Nature. 2013 Jul 11;499(7457):214-218. doi: 10.1038/nature12213. Epub 2013 Jun 16. PMID 23770567
- [Background] Leon-Castillo A, de Boer SM, Powell ME, Mileshkin LR, Mackay HJ, Leary A, Nijman HW, Singh N, Pollock PM, Bessette P, Fyles A, Haie-Meder C, Smit VTHBM, Edmondson RJ, Putter H, Kitchener HC, Crosbie EJ, de Bruyn M, Nout RA, Horeweg N, Creutzberg CL, Bosse T; TransPORTEC consortium. Molecular Classification of the PORTEC-3 Trial for High-Risk Endometrial Cancer: Impact on Prognosis and Benefit From Adjuvant Therapy. J Clin Oncol. 2020 Oct 10;38(29):3388-3397. doi: 10.1200/JCO.20.00549. Epub 2020 Aug 4. PMID 32749941
- [Background] Lu KH, Broaddus RR. Endometrial Cancer. N Engl J Med. 2020 Nov 19;383(21):2053-2064. doi: 10.1056/NEJMra1514010. No abstract available. PMID 33207095
- [Background] Mayakonda A, Lin DC, Assenov Y, Plass C, Koeffler HP. Maftools: efficient and comprehensive analysis of somatic variants in cancer. Genome Res. 2018 Nov;28(11):1747-1756. doi: 10.1101/gr.239244.118. Epub 2018 Oct 19. PMID 30341162
- [Background] McShane LM, Altman DG, Sauerbrei W, Taube SE, Gion M, Clark GM; Statistics Subcommittee of the NCI-EORTC Working Group on Cancer Diagnostics. Reporting recommendations for tumor marker prognostic studies (REMARK). J Natl Cancer Inst. 2005 Aug 17;97(16):1180-4. doi: 10.1093/jnci/dji237. PMID 16106022
- [Background] Meyer LA, Broaddus RR, Lu KH. Endometrial cancer and Lynch syndrome: clinical and pathologic considerations. Cancer Control. 2009 Jan;16(1):14-22. doi: 10.1177/107327480901600103. PMID 19078925
- [Background] Moore HM, Kelly AB, Jewell SD, McShane LM, Clark DP, Greenspan R, Hayes DF, Hainaut P, Kim P, Mansfield EA, Potapova O, Riegman P, Rubinstein Y, Seijo E, Somiari S, Watson P, Weier HU, Zhu C, Vaught J. Biospecimen reporting for improved study quality (BRISQ). Cancer Cytopathol. 2011 Apr 25;119(2):92-101. doi: 10.1002/cncy.20147. Epub 2011 Mar 22. PMID 21433001
- [Background] Onstad MA, Schmandt RE, Lu KH. Addressing the Role of Obesity in Endometrial Cancer Risk, Prevention, and Treatment. J Clin Oncol. 2016 Dec 10;34(35):4225-4230. doi: 10.1200/JCO.2016.69.4638. Epub 2016 Nov 7. PMID 27903150
- [Background] Orekoya O, Samson ME, Trivedi T, Vyas S, Steck SE. The Impact of Obesity on Surgical Outcome in Endometrial Cancer Patients: A Systematic Review. J Gynecol Surg. 2016 Jun 1;32(3):149-157. doi: 10.1089/gyn.2015.0114. PMID 27274182
- [Background] Raglan O, Kalliala I, Markozannes G, Cividini S, Gunter MJ, Nautiyal J, Gabra H, Paraskevaidis E, Martin-Hirsch P, Tsilidis KK, Kyrgiou M. Risk factors for endometrial cancer: An umbrella review of the literature. Int J Cancer. 2019 Oct 1;145(7):1719-1730. doi: 10.1002/ijc.31961. Epub 2019 Feb 20. PMID 30387875
- [Background] Seborova K, Koucka K, Spalenkova A, Holy P, Ehrlichova M, Sychra T, Chen L, Bendale H, Ojima I, Sandoval-Acuna C, Truksa J, Soucek P, Vaclavikova R. Anticancer regimens containing third generation taxanes SB-T-121605 and SB-T-121606 are highly effective in resistant ovarian carcinoma model. Front Pharmacol. 2022 Nov 9;13:971905. doi: 10.3389/fphar.2022.971905. eCollection 2022. PMID 36438837
- [Background] Seborova K, Hlavac V, Holy P, Bjorklund SS, Fleischer T, Rob L, Hruda M, Bouda J, Mrhalova M, Allah MMKAO, Vodicka P, Fiala O, Soucek P, Kristensen VN, Vodickova L, Vaclavikova R. Complex molecular profile of DNA repair genes in epithelial ovarian carcinoma patients with different sensitivity to platinum-based therapy. Front Oncol. 2022 Dec 2;12:1016958. doi: 10.3389/fonc.2022.1016958. eCollection 2022. PMID 36531044
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Vaclavikova R, Klajic J, Brynychova V, Elsnerova K, Alnaes GIG, Tost J, Kristensen VN, Rob L, Kodet R, Skapa P, Mrhalova M, Soucek P. Development of high-resolution melting analysis for ABCB1 promoter methylation: Clinical consequences in breast and ovarian carcinoma. Oncol Rep. 2019 Aug;42(2):763-774. doi: 10.3892/or.2019.7186. Epub 2019 Jun 5. PMID 31173253
- [Background] Vaclavikova R, Ehrlichova M, Hlavata I, Pecha V, Kozevnikovova R, Trnkova M, Adamek J, Edvardsen H, Kristensen VN, Gut I, Soucek P. Detection of frequent ABCB1 polymorphisms by high-resolution melting curve analysis and their effect on breast carcinoma prognosis. Clin Chem Lab Med. 2012 Nov;50(11):1999-2007. doi: 10.1515/cclm-2012-0103. PMID 23093106
- [Background] Walsh CS, Hacker KE, Secord AA, DeLair DF, McCourt C, Urban R. Molecular testing for endometrial cancer: An SGO clinical practice statement. Gynecol Oncol. 2023 Jan;168:48-55. doi: 10.1016/j.ygyno.2022.10.024. Epub 2022 Nov 15. PMID 36399812
- [Background] Wang S, Li H, Song M, Tao Z, Wu T, He Z, Zhao X, Wu K, Liu XS. Copy number signature analysis tool and its application in prostate cancer reveals distinct mutational processes and clinical outcomes. PLoS Genet. 2021 May 4;17(5):e1009557. doi: 10.1371/journal.pgen.1009557. eCollection 2021 May. PMID 33945534